CLINICAL TRIAL: NCT06788964
Title: A Phase 2 Study of Loncastuximab Tesirine and Rituximab as Bridging Therapy Prior to Standard-of-care CD19 CAR T-cell Therapy in Patients With Large B-cell Lymphoma
Brief Title: Loncastuximab Tesirine and Rituximab as Bridging Therapy Before Standard-of-care CAR-T Therapy in Patients With Large B-cell Lymphoma (CORAL)
Acronym: CORAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI184585
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Relapsed or Refractory Large B-cell Lymphoma
MeSH Terms: conditions — Recurrence | interventions — loncastuximab tesirine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: All Patients (Experimental): The study will investigate the effectiveness of Loncastuximab tesirine and Rituximab (Lonca-R) prior to standard of care CAR-T cell therapy.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Rituximab

INTERVENTIONS:
Drug: Loncastuximab Tesirine — Patients will receive Loncastuximab Tesirine intravenously for 1-6 cycles (every 21 days) prior to standard of care CAR-T cell therapy.
  Other Names: ZYNLONTA
Drug: Rituximab — Rituximab is administered intravenously for 1-6 cycles (every 21 days) prior to standard of care CAR-T cell therapy.
  Other Names: RITUXAN

SUMMARY:
The purpose of this clinical trial is to learn if the study treatment Loncastuximab tesirine and Rituximab is safe and efficient before standard of care chimeric antigen receptor T-cell (CAR-T) therapy in patients with relapsed or refractory large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥ 18 years.
* Intended to receive commercial CD19-directed CAR-T cell therapy (axi-cel and liso-cel).
* Need for bridging therapy as deemed clinically necessary by the treating physician.
* Relapsed or refractory DLBCL, tFL or PMBCL as defined by the 2016 World Health Organization classification (including patients with DLBCL transformed from indolent lymphoma), or high-grade B-cell lymphoma (HGBL), not otherwise specified, and HGBL with MYC and BCL2 and/or BCL6 rearrangements.

  --Relapsed (disease that has recurred following a response) or refractory (disease that failed to respond to prior therapy) disease following at least one multi-agent systemic treatment regimen.
* Measurable disease as defined by the 2014 Lugano Classification as assessed by positron-emission tomography (PET)- computed tomography (CT) or by CT or magnetic resonance imaging (MRI) if the tumor is not fluorodeoxyglucose (FDG)-avid on screening PET-CT.
* ECOG Performance Status ≤ 2.
* Time between prior anticancer therapy and first dose of lonca-R as below

  * Autologous hematopoietic cell transplantation - At least 30 days
  * Allogeneic hematopoietic cell transplantation - At least 60 days
  * Cytotoxic chemotherapy - At least 21 days
  * Non-cytotoxic chemotherapy (e.g., small molecule inhibitor) - At least 14 days
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count (ANC) ≥ 1000/mm3
    * Platelet count ≥ 75,000/mm3
    * Hemoglobin ≥ 8 g/dL
  * Hepatic:

    * Bilirubin ≤1.5 x upper limit of normal (ULN) or ≤3 x ULN with document liver involvement and/ or Gilbert's disease
    * Transaminases (AST or ALT) ≤ 3 x ULN or ≤ 5 x ULN with documented liver involvement
  * Renal:

    * Estimated creatinine clearance ≥ 60 mL/min by Cockcroft-Gault formula.
* For female subjects: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
    * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or
    * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Female subjects of childbearing potential and male subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception and the lactation requirements as described in Sections 5.41.1 and 5.4.2.
* Subjects or their legal representatives must be able to read, understand, and provide informed consent to participate in the trial.
* Willing and capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol

Exclusion Criteria:

* Previous treatment with any anti-CD19 therapy including lonca or prior CD19 CAR T-cell therapy
* Subjects receiving investigational CAR-T products
* Major surgery within 4 weeks prior to starting study therapy.
* History of bleeding diathesis (e.g., von Willebrand's disease), hemophilia, or active bleeding.
* Subjects with chronic liver disease with hepatic impairment Child-Pugh class C
* Pregnant or lactating or intending to become pregnant during the study
* Active graft-versus-host disease
* Post-transplantation lymphoproliferative disorders
* Active autoimmune disease which, in the opinion of the investigator, may negatively impact subject safety or interfere with study participation.
* The diagnosis of another malignancy which, in the opinion of the investigator, is likely to negatively impact subject safety or interfere with study participation.
* Subjects with known CNS involvement.
* Significant medical diseases or conditions including those requiring substantial changes in concomitant medications, as assessed by the investigator, that would substantially increase the risk-to-benefit ratio of participating in the study. This includes, but is not limited to the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class III or IV, unstable angina pectoris, serious cardiac arrhythmias.
    * Myocardial infarction (MI) within 6 months before the first dose.
    * QTc prolongation defined as a QTcF > 480 ms.
    * Congenital long QT syndrome or a corrected QT measure (QTc) interval of >480 ms at screening (unless secondary to pacemaker or bundle branch block).
  * Severe pulmonary disease
  * Uncontrolled diabetes mellitus
  * Severely immunocompromised state
  * Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Active systemic bacterial, viral, fungal, or other infection requiring systemic treatment at time of screening
* HIV infection.
* Subjects with evidence of active hepatitis B infection, based on positive surface antigen or Hepatitis B DNA PCR are excluded. Subjects who are Hepatitis B core antibody positive must take prophylaxis with entecavir or equivalent and be willing to undergo monthly Hepatitis B DNA PCR testing. Subjects with active Hep C patients may be enrolled if other parameters precluding hepatic impairment are met and they are not undergoing active therapy for hepatitis C.
* Known prior severe hypersensitivity to a CD19 antibody, lonca (including SG3249) or any of its excipients, or history of positive serum human ADA to a CD19 antibody.
* Subjects taking prohibited medications as described in Section 6.8.1. A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
The complete response (CR) rate at D30 post CAR-T(+/- 7 days) post CAR-T administration per Lugano 2014 criteria. | 1 month
  To evaluate the efficacy of SOC CAR T-cell therapy in patients with R/R large B-cell lymphoma following bridging with lonca-R.
Duration of cytopenias post CAR-T (as defined by the NIH CTCAE, version 5.0) D30 post CAR-T (+/- 7 days). | 1 month
  To evaluate toxicities post CAR-T
Severity of cytopenias post CAR-T (as defined by the NIH CTCAE, version 5.0) D30 (+/- 7 days). | 1 month
  To evaluate toxicities post CAR-T
Rate of infections D30 (+/- 7 days). | 1 month
  To evaluate toxicities post CAR-T

SECONDARY OUTCOMES:
CD19 expression as measured by flow cytometry and IHC on biopsies obtained pre- and post-lonca-R (optional) and post-CAR-T (optional but strongly recommended) | 5 years
  To determine whether CD19 expression is reduced in patients who receive bridging with lonca-R prior to CAR-T.
ORR defined as the proportion of subjects achieving a confirmed PR or CR at D30 (+/- 7 days) post CAR-T per Lugano 2014 criteria1. | 1 month
  To evaluate the level of disease control provided by bridging lonca-R
Best response rate per Lugano 2014 criteria following CAR-T (based on imaging up until D90 post CAR-T) | 3 months
  To evaluate the level of disease control provided by bridging lonca-R
ORR defined as the proportion of subjects achieving a confirmed PR or CR post lonca-R (pre-CAR-T) | 5 years
  To evaluate the level of disease control provided by bridging lonca-R
Level of disease control (measured as percentage) with lonca-R as evaluated by CT measurements and metabolic tumor volume on PET pre and post Lonca-R | 5 years
  To evaluate the level of disease control provided by bridging lonca-R
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by severity (as defined by the NIH CTCAE, version 5.0) | 5 years
  To assess the safety and tolerability of lonca-R in the study population.
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by seriousness. | 5 years
  To assess the safety and tolerability of lonca-R in the study population.
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by duration. | 5 years
  To assess the safety and tolerability of lonca-R in the study population.
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by relationship to study treatment. | 5 years
  To assess the safety and tolerability of lonca-R in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Narendranath Epperla, MD, MS, FACP, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No